CLINICAL TRIAL: NCT03494738
Title: Development of an Epigenetic Biomarker for Prediction of Fetal Alcohol Spectrum Disorder
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CAMC Health System (Other)
Collaborators: United States Drug Testing Laboratories, Inc. (Unknown)
Responsible Party: Principal Investigator, Stefan Maxwell, Medical Director of NICU, CAMC Women and Children's Hospital, CAMC Health System
Other Study IDs: 17-388
Record Dates: First submitted 2018-03-23; First posted 2018-04-11 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Fetal Alcohol Spectrum Disorders
Keywords: Prenatal alcohol exposure
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dried bloodspots obtained from umbilical cord at birth and heel sticks at 24-48 hours post birth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newborn infants: Neonates born from consented women at the study hospital

SUMMARY:
The objective of the study is to validate epigenetic changes as biomarkers in a prospective sampling of newborn blood samples collected at birth (umbilical cord blood) and during routine screening (heel stick blood) in newborns concurrently tested for alcohol exposure levels by PEth blood spot testing.

DETAILED DESCRIPTION:
Fetal alcohol spectrum disorders (FASD) are a group of conditions that can occur in a person whose birth mother consumed alcohol during pregnancy. The effects can include physical problems and/or difficulties with behavior and learning. When clinicians identify FASD early, intervention approaches can minimize the potential impact and lessen or even prevent disabilities. Thus, objective markers for prenatal alcohol exposure are desired.

Using dried blood spots from the umbilical cord and a heel stick of newborns, this study will use Phosphatidylethanol (PEth), a novel biomarker for alcohol exposure, to identify and characterize infants' exposure to alcohol before birth. Additionally, the dried blood spots will used to validate the use of screening assays using epigenetic changes as markers for prenatal alcohol exposure. Epigenetic changes are heritable changes in DNA that affect DNA function but do not change DNA sequence. The use of PEth testing will allow for the correlation of prenatal alcohol exposure levels with epigenetic changes. Women will be consented prior to delivery for participation in this prospective study. The study will be conducted in collaboration with United States Drug Testing Laboratories, Inc. (USDTL).

ELIGIBILITY:
Women:

Inclusion criteria

* Women aged ≥ 18 years and currently pregnant at time of enrollment
* Women who plan to and then deliver their infants at CAMC Women and Children's Hospital

Exclusion criteria

* Women aged < 18 years
* Women not pregnant
* Women who do not plan to deliver or did not end up delivering their infants at CAMC Women and Children's Hospital

Infants:

Inclusion criteria

* Birth mother was consented prior to delivery
* Live birth at CAMC Women and Children's Hospital

Exclusion criteria

* Birth mother was NOT consented prior to delivery
* Stillborn

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women will be consented for study participation of their neonates prior to delivery.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Epigenetic changes as biomarkers of prenatal alcohol exposure | 48 hours post birth
  Validation of the epigenetic changes as biomarkers of newborn blood samples collected at birth (umbilical cord blood) and during routine screening (heel stick blood) in newborns concurrently tested for alcohol exposure levels by PEth blood spot testing.

SECONDARY OUTCOMES:
Optimal timing to obtain samples from neonates for prenatal alcohol detection | 48 hours post birth
  To compare PEth levels and epigenetic changes in dried blood spots obtained via umbilical cord at birth verses heel stick at 48 hours post-birth.

OTHER OUTCOMES:
Gestational age at birth | at birth
Small for gestational age: composite of small for gestational age (<10% percentile) for weight or length or head circumference | at birth
Postnatal complications: Composite of having one or more of the following: neonatal sepsis, necrotizing enterocolitis, respiratory distress syndrome, hyperbilirubinemia, intraventricular hemorrhage | 28 days post birth

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Maxwell, MD, Principal Investigator — CAMC Women and Children's Hospital
Locations (1):
- CAMC - Women and Children's Hospital, Charleston, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No